CLINICAL TRIAL: NCT01525511
Title: Open-Label Study to Evaluate Potential Pharmacokinetic Interaction of Orally Administered Primaquine and Dihydroartemisinin-Piperaquine in Healthy Adult Subjects
Brief Title: Pharmacokinetic Study of Primaquine and Dihydroartemisinin-Piperaquine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FTM1102
Record Dates: First submitted 2012-01-16; First posted 2012-02-03 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Primaquine only followed by Dihydroartemisinin-piperaquine and followed by Primaquine together with Dihydroartemisinin-piperaquine.
  Interventions: Drug: A
- Group B (Active Comparator): Primaquine only followed by Primaquine together Dihydroartemisinin-piperaquine and followed by Dihydroartemisinin-piperaquine only.
  Interventions: Drug: B

INTERVENTIONS:
Drug: A — Subject will receive primaquine (PQ) then receive dihydroartemisinin-piperaquine (DHA-PQP)after 1 week washout period and receive PQ together with DHA-PQP for the third regimen after 8 weeks washout period.
  Primaquine:
  * 1 tablet of primaquine phosphate contains: 26.3 mg (15 mg base)
  * Dosage: 2 tablets
  DHA-PQP:
  * 1 tablet of Eurartesim contains: DHA 40 mg: piperaquine 320 mg
  * Dosage: 3 tablets
  Arms: Group A
Drug: B — Subject will receive primaquine (PQ) then receive PQ together dihydroartemisinin-piperaquine (DHA-PQP) after 1 week washout period and receive DHA-PQP for the third regimen after 8 weeks washout period.
  Primaquine:
  * 1 tablet of primaquine phosphate contains: 26.3 mg (15 mg base)
  * Dosage: 2 tablets
  DHA-PQP:
  * 1 tablet of Eurartesim contains: DHA 40 mg: piperaquine 320 mg
  * Dosage: 3 tablets
  Arms: Group B

SUMMARY:
The observed changes of P. falciparum sensitivity to artemisinin leads to the intensification of early detection as well as treatment monitoring in malaria infection. It is widely accepted that the development of resistance can be delayed by the use of combination therapy, especially artemisinin-based combination therapies (ACTs). The resistance problem is considered extremely serious and as the consequence WHO has recommended that all monotherapy for malaria should be stopped Current WHO guideline recommends the drug combination regimens using ACT with effective partner medicines to decrease the risk of development or spreading of artemisinin resistance.

Dihydroartemisinin-piperaquine (DHA-PQP); the fixed-dose combination of Dihydroartemisinin (DHA) and Piperaquine phosphate (PQP) is now one of the recommended drugs by WHO as the oral treatment for uncomplicated P. falciparum. DHA-PQP composes of both blood schizonticidal drugs, with different mechanism of action and different half-life to improve the therapeutic efficacy and to prevent the development of drug resistance to the individual drug. Moreover, it is beneficial for the mutual protection against resistance and long lasting protection against new infection, due to long half-life of PQP.

Primaquine is an effective gametocytocidal for P. falciparum transmission prevention and as tissue killing for the radical cure in Plasmodium vivax and Plasmodium ovale infection. It will be given only in the presence of other antimalarials, so it is necessary that the data of the potential drugs interaction of primaquine and DHA-PQP should be characterized. It is inevitable that in the near future, Dihydroartemisinin-piperaquine (DHA-PQP) and primaquine combination treatment becomes necessary. These drugs are metabolized by cytochrome P450 enzyme which potentially causes pharmacokinetic alteration, resulting in clinically significant drug-drug interactions that can cause unanticipated adverse reactions or therapeutic failures because of the suboptimal exposure of the parasite.

This study is planned to evaluate potential pharmacokinetic interaction of orally administered primaquine (PQ) and dihydroartemisinin-piperaquine (DHA-PQP) in healthy adult subjects. The results of these interaction studies are important in order to provide clinical guidance for the optimum combination of primaquine and DHA-PQP treatment regimens in malaria infections.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination.
2. Males and Females non-smoker aged between 18 years to 60 years.
3. Males and Females weight between 36-75 kilograms.
4. A female is eligible to enter and participate in this study if she is:

   * of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy
   * or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
   * or of childbearing potential, has a negative serum pregnancy test at screening and prior to start the study drug in each period, and abstain from sexual intercourse or agrees to using effective contraceptive methods (e.g., intrauterine device, hormonal contraceptive drug, tubal ligation or female barrier method with spermicide) during the study until completion of the follow-up procedures
5. A male is eligible to enter and participate in this study if he: agrees to abstain from (or use a condom during) sexual intercourse with females of childbearing potential or lactating females; or is willing to use a condom/spermicide, during the study until completion of the follow-up procedures.
6. Provide a signed and dated written informed consent prior to study participation.
7. Normal electrocardiogram (ECG) with QTc <450 msec.
8. Willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. The subject has evidence of active substance abuse that may compromise safety, pharmacokinetics, or ability to adhere with protocol instructions.
3. A positive pre-study hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
4. Subjects with a personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de points (heart failure, hypokalemia) or with a family history of sudden cardiac death.
5. A creatinine clearance <70 mL/min as determined by Cockcroft-Gault equation:

   CLcr (mL/min) = (140 - age) * Wt / (72 * Scr) (multiply answer by 0.85 for females) Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dL [Cockcroft, 1976].
6. History of alcohol or substance abuse or dependence within 6 months of the study.
7. Use of prescription or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 times the drug half-life (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety; the investigator will take advice from the manufacturer representative as necessary.
8. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half life, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
9. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample during each regimen.
10. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period. Note: This does not include plasma donation.
11. Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
12. Lack of suitability for participation in this study, including but not limited to, unstable medical conditions, systemic disease manifested by tendency to granulocytopenia e.g. rheumatoid arthritis and lupus erythematosus that in the opinion of the investigator would compromise their participation in the trial.
13. AST or ALT >1.5 upper limit of normal (ULN)
14. Subjects with history of renal disease, hepatic disease, and/or cholecystectomy
15. G6PD deficient detected by Beutler's dye test.
16. Abnormal methaemoglobin level.
17. History of antimalarial drugs use including but not limited to mefloquine, chloroquine, primaquine, artesunate, piperaquine and pyronaridine treatment within 12 months.
18. Subject who received quinacrine in last 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) for Primaquine | 36 days
  Area under the concentration-time curve [(AUC(0-∞) and AUC(0-last)] and maximal concentration (Cmax) for primaquine and metabolites when given alone or together with DHA-PQP.
Area Under Curve (AUC) for Dihydroartemisinin (DHA) and Piperaquine (PQP) | 36 days
  Area under the concentration-time curve [(AUC(0-∞) and AUC(0-last)] and maximal concentration (Cmax) for piperaquine and dihydroartemisinin when given alone as DHA-PQP or together with primaquine.

SECONDARY OUTCOMES:
Clearance rate and half life of Primaquine and its metabolites | 36 days
  Primaquine, carboxyprimaquine (and other detectable major metabolites) elimination clearance rate (CL/F), terminal elimination half-life (t1/2) and apparent volume of distribution (Vd) Dihydroartemisinin and piperaquine elimination clearance rate (CL/F), terminal elimination half-life (t1/2) and apparent volume of distribution (Vd).
Safety of Dihydroartemisinin-Piperaquine (DHA-PQP) | 36 days
  Safety and tolerability parameters, including adverse events, clinical laboratory, and vital signs assessments, in particular QTc prolongation for DHA-PQP
Pharmacogenetic polymorphisms | 36 days
  Pharmacogenetic polymorphisms in the case of unusually high or low drug levels.

CONTACTS AND LOCATIONS:
Overall Officials: Sasithon Pukrittayakamee, MD, Principal Investigator — Mahidol University
Locations (1):
- Hospital of Tropical Diseases, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Derived] Hanboonkunupakarn B, Ashley EA, Jittamala P, Tarning J, Pukrittayakamee S, Hanpithakpong W, Chotsiri P, Wattanakul T, Panapipat S, Lee SJ, Day NP, White NJ. Open-label crossover study of primaquine and dihydroartemisinin-piperaquine pharmacokinetics in healthy adult thai subjects. Antimicrob Agents Chemother. 2014 Dec;58(12):7340-6. doi: 10.1128/AAC.03704-14. Epub 2014 Sep 29. PMID 25267661